CLINICAL TRIAL: NCT06746753
Title: Dysfunctional Renin-Angiotensin System in Septic Shock
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00115287; 11773 (Other: National Heart. Lung, and Blood)
Record Dates: First submitted 2024-12-18; First posted 2024-12-24 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Septic Shock
Keywords: sepsis; kidney disease; intensive care
MeSH Terms: conditions — Shock, Septic; Sepsis; Kidney Diseases | interventions — Angiotensin II; Norepinephrine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Angiotensin II (Experimental): Continuous infusion of Angiotensin II for up to 48 hours
  Interventions: Drug: Angiotensin II
- Norepinephrine (Active Comparator): Continuous infusion of Norepinephrine for up to 48 hours
  Interventions: Drug: Norepinephrine

INTERVENTIONS:
Drug: Angiotensin II — randomized to receive Angiotensin II continuous infusion for up to 48 hours
  Arms: Angiotensin II
Drug: Norepinephrine — randomized to receive Norepinephrine continuous infusion for up to 48 hours
  Arms: Norepinephrine

SUMMARY:
Despite best therapy efforts, sepsis and septic shock are associated with mortality rates of up to 40%. This clinical trial will determine the benefit of exogenous Angiotensin II versus norepinephrine (conventional care) treatment in septic shock patients. This trial will determine whether there are better predictors of septic shock severity. This approach may inform more appropriate treatment regimens and improve outcomes for these patients.

DETAILED DESCRIPTION:
This study will determine whether normalization of renin-angiotensin-aldosterone system (RAAS) signaling in sepsis occurs more rapidly with treatment with Angiotensin II compared with conventional vasopressors. Trial samples will be used to identify the best RAAS biomarker predictor of treatment response via in-depth longitudinal analysis of RAAS component and to determine the extent and mechanisms of Angiotensin II impact on innate immune function during sepsis. Successful accomplishment of our aims will provide the capability to improve endotyping of septic patients by establishing the most precise and robust measurement of renin (and RAAS dysfunction). This work will improve staging and clinical precision and will facilitate the criteria for therapeutic development of targets in septic shock.

ELIGIBILITY:
Inclusion Criteria:

* The presence of septic shock, defined by sepsis-3 criteria
* The requirement for Norepinephrine of at least 10 micrograms/minute up to 35 micrograms/minute for at least 1 hour, with or without Vasopressin, to maintain a mean arterial pressure of 65 mmHg
* Clinical suspicion or proven evidence of infection

Exclusion Criteria:

* Age <18 years
* Prisoners
* Pregnant women
* Patients for whom urgent surgery is anticipated
* Leukocyte count <1,000 cells/μL
* Absolute monocyte count <200 cells/μL
* Bone marrow transplant within the past 30 days
* Patients that will be withdrawing aggressive resuscitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-07 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Mean Renin Level - Hour 24 | Hour 24
  Mean renin level as a measure of renin-angiotensin-aldosterone system restoration. Normal levels of active renin <1.1 pM (40 pg/mL). A level higher than normal can indicate level of shock.

SECONDARY OUTCOMES:
Norepinephrine Equivalent Dose Requirement (NEE) | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  NEE indicates severity of shock and need for vasopressors to support blood pressure. Normal range is 0.0-1.0 mcg/kg/min. Levels above normal indicate shock and need for vasopressors. The higher the level the more severe.
Number of Days Without Renal Replacement Therapy | Day 28
  Number of days without renal replacement therapy
Number of Days of Vasopressor Use | Day 28
  Number of days without vasopressor use
Number of Days Without Mechanical Ventilation | Day 28
  Number of days without invasive mechanical ventilation
Number of Hours Vasopressor Free | Hour 72
  Number of hours without requiring vasopressors during first 72 hours after randomization
Number of Hours Alive | Hour 72
  Number of hours alive during first 72 hours after randomization
Number of Days Alive | Day 28
  Number of days alive
Mean Renin Level | Baseline, Hour 3, Hour 12, Hour 48
  Mean renin level as a measure of renin-angiotensin-aldosterone system restoration. Normal levels of active renin <1.1 pM (40 pg/mL). A level higher than normal can indicate level of shock.
Sequential Organ Failure Assessment (SOFA) Score | Baseline, Hour 24, Hour 48
  SOFA score indicates the number and severity of failed organs and provides prognostic information on in-hospital survival in patients with severe sepsis and septic shock. Score above 0 indicates organ failure. The higher the score the more failed organs and degree of organ failure.
APACHE-II Score | Baseline, Hour 24, Hour 48
  APACHE-II score assesses severity of illness in critically ill patients and indicates risk of mortality. Score range 0-10 low risk of mortality, 11-20 moderate risk, 21-30 high risk, 31 or above very high risk.
Lactate Level | Baseline, Hour 3, Hour 12, Hour 48
  Lactate is an indicator of sepsis severity. Levels 2.3-20 mmol/L indicate sepsis. The higher the score the more severe.
Kidney Disease Improving Global Outcomes (KDIGO) Stage | Baseline, Hour 24, Hour 48
  Participant stage of acute kidney injury will be determined as follows Stage 1: Increase in serum creatinine ≥ 0.3 mg/dL in 48 hours or 1.5 to 1.9 multiplied by baseline (in 7 days); Stage 2: 2.0 to 2.9 multiplied by baseline serum creatinine; Stage 3: 3.0 or more multiplied by baseline; increase in serum creatinine ≥ 4.0 mg/dL; or beginning of renal replacement therapy regardless of a previous KDIGO stage. Higher stage indicates higher severity of renal failure.
Creatinine Level | Baseline, Hour 24, Hour 48
  Creatinine level is an indicator of renal disease severity. Normal range for women 0.7-1.3 mg/dL, men 0.6-1.1 mg/dL. Levels higher than normal indicate renal disease. The higher the level the more severe.
BUN Level | Baseline, Hour 24, Hour 48
  BUN level is an indicator of renal disease severity. Levels above 24 mg/dL indicate renal disease. The higher the level the more severe.
Bicarbonate Level | Baseline, Hour 24, Hour 48
  Bicarbonate level is an indicator of acid base disturbance severity. Normal range is 22-29 mEq/L. Levels above or below the normal range indicate acid base disturbance. The higher the score the more severe.
Number of Participants with Acute Respiratory Distress Syndrome (ARDS) | Baseline, Hour 24, Hour 48
  Number of participants with ARDS
SpO2/FiO2 Ratio Level | Baseline, Hour 24, Hour 48
  SpO2/FiO2 ratio level is an indicator of lung injury severity. Mild severity 315-235, moderate severity 148-235, severe <148.
PaO2/FiO2 Ratio Level | Baseline, Hour 24, Hour 48
  PaO2/FiO2 ratio level is an indicator of lung injury severity. Mild severity 201-300 mmHg; moderate severity 101-200 mmHg, severe ≤ 100 mmHg.
Serum Aspartate Aminotransferases Level | Baseline, Hour 24, Hour 48
  Serum aspartate aminotransferases level is an indicator of liver injury severity. Normal range 8-48 U/L. Levels above normal indicate livery injury. The higher the level the more severe.
Alanine Aminotransferases Level | Baseline, Hour 24, Hour 48
  Alanine aminotransferases level is indicator of liver injury severity. Normal range 7-55 U/L. Levels higher than normal indicate liver injury. The higher the level the more severe.
Alkaline Phosphatase Level | Baseline, Hour 24, Hour 48
  Alkaline phosphatase level is an indicator of liver injury severity. Normal range 40-129 U/L. Levels higher than normal indicate liver injury. The higher the level the more severe.
Bilirubin Level | Baseline, Hour 24, Hour 48
  Bilirubin level is an indicator of liver injury severity. Normal range 0.1-1.2 mg/dL. Levels higher than normal indicate liver injury. The higher the liver the more severe.
Albumin Level | Baseline, Hour 24, Hour 48
  Albumin level is an indicator of liver injury severity. Normal range 3.5-5.0 g/dL. Levels higher than normal indicate liver injury. The higher the level the more severe.
Troponin I Level | Baseline, Hour 24, Hour 48
  Troponin I level is an indicator of cardiac myocyte injury. Normal range 0-0.04 ng/mL. Levels higher than normal indicate cardiac myocyte injury. The higher the level the more severe.
Troponin T Level | Baseline, Hour 24, Hour 48
  Troponin T level is an indicator of cardiac myocyte injury. Normal range 0-0.01 ng/mL. Levels higher than normal indicate cardiac myocyte injury. The higher the level the more severe.
Neutrophil Gelatinase-Associated Lipocalin Serum Level | Baseline, Hour 24, Hour 48
  Neutrophil gelatinase-associated lipocalin serum level indicates risk of kidney injury. Normal serum level is <10 mcg/L. Levels higher than normal indicate risk of kidney injury.
Neutrophil Gelatinase-Associated Lipocalin Urine Level | Baseline, Hour 24, Hour 48
  Neutrophil gelatinase-associated lipocalin urine level indicates risk of kidney injury. Normal urine level is ≤50 ng/ml. Risk of kidney disease: Low risk 51-149 ng/ml, moderate risk 150-299 ng/ml, and high risk ≥300 ng/ml.
Kidney Injury Molecule-I Urine Level | Baseline, Hour 24, Hour 48
  Kidney injury molecule-I urine level is used to detect kidney injury. Normal level is <1 ng/ml. Levels higher than normal indicate ischemic kidney injury.
Kidney Injury Molecule-I Blood Level | Baseline, Hour 24, Hour 48
  Kidney injury molecule-I blood level is used to detect kidney injury. Normal levels 0.42-2.0 ng/ml. Levels higher than normal indicate kidney injury. The higher the level the more severe.
Soluble Receptor for Advanced Glycation End Product Level | Baseline, Hour 24, Hour 48
  Soluble receptor for advanced glycation end product level is a marker of aging, hypertension and diabetes. Normal range is 647-1248 pg/ml. Levels higher than normal indicate risk for hypertension and diabetes.
Angiopoietin-2 Level | Baseline, Hour 24, Hour 48
  Angiopoietin-2 level is a marker of inflammation. Normal range is 1434-4141 pg/mL. Levels higher than normal indicate inflammation.
Syndecan-1 Level | Baseline, Hour 24, Hour 48
  Syndecan-1 level is a marker of disease severity in critically ill patients. Levels >20ng/ml indicate severe disease. The higher the level the more severe.
Protein C Level | Baseline, Hour 24, Hour 48
  Protein C level is an indicator of inflammation and thrombotic state. Normal level is <8 mg/L. Levels higher than normal indicate inflammation and thrombotic state. The higher the level the more severe.
Neuron-Specific Enolase Level | Baseline, Hour 24, Hour 48
  Neuron-specific enolase level is an indicator of brain injury. Normal range is 16-17 ug/L. Levels higher than normal indicate brain injury. The higher the level the more severe.
S-100β Level | Baseline, Hour 24, Hour 48
  S-100β level is indicator of brain injury. Normal range is 0.02-0.05 μg/dL. Levels higher than normal indicate brain injury. The higher the number the more severe.
TNFα Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  TNFα level is an indicator of systemic inflammation. Normal levels are 75 +/- 15 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
sTNFR1 Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  sTNFR1 level is an indicator of systemic inflammation. Normal levels are <2.4 ng/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
IL-6 Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  IL-6 level is an indicator of systemic inflammation. Normal range is 0-43.5 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
sIL-6R Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  sIL-6R level is an indicator of systemic inflammation. Normal range is 14-46 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
IL-8 Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  IL-8 level is an indicator of systemic inflammation. Normal range is 0-66.1 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
IL-1β Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  IL-1β level is an indicator of systemic inflammation. Normal range is 0.5-12 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
Interferon Gamma Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  IFN-ɣ level is an indicator of systemic inflammation. Normal range is 0-8.6 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
IL12p70 Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  IL12p70 level is an indicator of systemic inflammation. Normal range is 0-1.9 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
IL-17 Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  IL-17 level is an indicator of systemic inflammation. Normal range is 0-1.4 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
MIP1-alpha Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  MIP1-αlpha level is an indicator of systemic inflammation. Normal range is 0-208 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
MIP1-beta Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  MIP1-beta level is an indicator of systemic inflammation. Normal range is 59-647 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
IP-10 Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  IP-10 level is an indicator of systemic inflammation. Normal range is 4.8-9.8 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
IL-10 Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  IL-10 level is an indicator of systemic inflammation. Normal range is 4.8-9.8 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
IL-1RA Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  IL-1RA level is an indicator of systemic inflammation. Normal range is 100-300 ng/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
IL-12p40 Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  IL-12p40 level is an indicator of systemic inflammation. Normal range is 0.064-1000 pg/ml. Levels higher than normal indicate inflammation. The higher the score the more severe.
C reactive protein (CRP) Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  CRP level is an indicator of systemic inflammation. Normal range is 0-10 mg/dl. Levels higher than normal indicate inflammation. The higher the score the more severe.
Procalcitonin Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  Procalcitonin level is an indicator of systemic inflammation. Levels >0.25 mg/ml indicate inflammation and infection. The higher the score the more severe.
Platelet Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  Platelet level is an indicator of systemic inflammation and thrombocytosis. Normal range is 150000-450000 platelets per microliter. Levels higher than normal indicate inflammation and thrombocytosis. The higher the score the more severe.
Absolute Neutrophil Count Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  Absolute neutrophil count level is an indicator of inflammation and infection/sepsis. Normal range is 2500-7000 neutrophils per microliter. Levels higher than normal indicate inflammation, infection/sepsis. The higher the score the more severe.
Absolute Granulocyte Count Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  Absolute granulocyte count level is an indicator of inflammation and infection/sepsis. Normal range is 1500-8500 granulocytes per microliter. Levels higher than normal indicate inflammation, infection/sepsis. The higher the score the more severe.
Absolute Lymphocytes Count Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  Absolute lymphocyte count level is an indicator of inflammation and infection/sepsis. Normal range is 1000-4800 granulocytes per microliter. Levels higher than normal indicate inflammation, infection/sepsis. The higher the score the more severe.
Neutrophil-Lymphocyte Ratio Level | Baseline, Hour 3, Hour 12, Hour 24, Hour 48
  Neutrophil-lymphocyte ratio level is an indicator of inflammation and infection/sepsis or marrow malignancy. Normal range is 1-2. Levels higher than normal indicate inflammation, infection/sepsis, marrow malignancy. The higher the score the more severe.

OTHER OUTCOMES:
Patients with New Deep Venous Thrombosis | Day 28
  Number of patients with development of new deep venous thrombosis
Patients with New Pulmonary Embolism | Day 28
  Number of patients with development of new pulmonary embolism
Patients with New-Onset Atrial Fibrillation | Hour 72
  Number of patients with new-onset atrial fibrillation
Patients with New-Onset Ventricular Arrhythmias | Hour 72
  Number of patients with new-onset ventricular arrhythmias

CONTACTS AND LOCATIONS:
Overall Officials: Ashish Khanna, MD, Principal Investigator — Atrium Health Wake Forest Baptist
Locations (1):
- Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No